CLINICAL TRIAL: NCT02388932
Title: Phase I Dose Escalation Study of Stereotactic Body Radiotherapy for Carcinoma of the Head and Neck in High Risk Patients Who Are Ineligible/Refuse Standard of Care Therapy
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With High Risk Locally Advanced Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8314; NCI-2014-02279 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE8314; CASE 8314 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Recurrent Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage II Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage III Hypopharyngeal Squamous Cell Carcinoma; Stage III Laryngeal Squamous Cell Carcinoma; Stage III Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage III Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage III Oral Cavity Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IVA Hypopharyngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IVA Oral Cavity Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Hypopharyngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Squamous Cell Carcinoma; Stage IVB Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IVB Oral Cavity Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Hypopharyngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Squamous Cell Carcinoma; Stage IVC Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IVC Oral Cavity Squamous Cell Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiosurgery; Positron-Emission Tomography; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (SBRT) (Experimental): Participants undergo Stereotactic Body Radiation Therapy in 5 fractions at least 40 hours apart over 10-18 days.
  Three dose levels: 40Gy and 45Gy all in 5 fractions. Each initial dose level will have 6 participants allocated to them. All participants are assessed at their 3 month post SBRT visit for Dose-Limiting Toxicities (DLTs). If ≤1 participant experiences a DLT, participants will be enrolled at the next dose level. If ≥3 participants experience a DLT, further accrual will be permanently halted and the study stopped. If 2 participants experience a DLT, then an additional 6 participants will be enrolled at the same dose level. In this setting, if ≤ 3/12 participants have a DLT, participants will be enrolled at the next dose level. If ≥ 4/12 participants have a DLT, further accrual will be permanently halted and the study stopped and 35 Gy will not be recommended as safe.
  The dosing strategy for the 2nd (45Gy) cohort will be identical to the first.
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Device: Positron Emission Tomography; Device: Computed Tomography; Other: Quality-of-Life Assessment

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT
Device: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan
Device: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; CT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I trial studies the side effects and best dose of stereotactic body radiation therapy (SBRT) in treating participants with head and neck cancer that has spread from where it started to nearby tissue or lymph nodes and is at high risk for continuing to spread because the participant cannot undergo standard chemotherapy. Stereotactic body radiation therapy is a specialized radiation therapy that delivers radiation directly to the tumor in smaller doses over several days, which may kill more tumor cells and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the maximum tolerated dose of head and neck stereotactic body radiation therapy (SBRT) in a high risk participant population ineligible for standard chemoradiotherapy.

SECONDARY OBJECTIVES:

I. Assess profiles of SBRT toxicity and examine participant (including co-morbidities), tumor and treatment related factors that are associated with SBRT related toxicity.

II. Identify any dose volume parameters that are associated with SBRT related toxicity.

III. Explore potential dose response relationships between higher SBRT dosing and radiographic response.

IV. Assess impact of SBRT on participants' quality of life.

OUTLINE: This is a dose-escalation study.

Participants undergo SBRT in 5 fractions at least 40 hours apart over 10-18 days.

After completion of study treatment, participants are followed up at 0.5, 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have squamous cell carcinoma proven by histologic diagnosis; for cancers of the oropharynx, p16 staining by immunohistochemistry must be negative; for cancers of the larynx, hypopharynx, oral cavity, nasopharynx, paranasal sinuses, p16 staining is not required
* The participant must have clinical stage T1-4, N0-3, M0-1, stage II-IVC carcinoma as per the 7th edition of the American Joint Committee on Cancer (AJCC) staging manual; participants with T1N0M0 will be ineligible; participants with metastatic disease with a limited metastatic burden are eligible if obtaining local control is determined by their treating oncologist to be an important therapeutic goal
* The participant must have imaging documenting a primary tumor, or involved lymph node, ≥ 2.5 cm in greatest dimension
* PET/CT is required for all participants, unless contraindicated; this may be acquired prior to study entry or after enrollment prior to SBRT planning
* The participant must have a history and physical documented within four weeks of registration and be deemed by a medical oncologist to be ineligible for standard continuous course chemoradiotherapy with cisplatin
* Karnofsky performance status (PS) ≥ 40
* Female participants cannot be of childbearing age, or if they are, must have a negative pregnancy test prior to enrollment and be willing to use contraceptives during treatment and continue for 6 additional months
* Participants must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants with T1N0M0 stage I disease
* Participants who are receiving any other investigational agents
* Participants with non-squamous cell histology
* Participants with life expectancy < 6 months
* Participants who cannot lie flat for 20 minutes
* Participants with prior history of head and neck radiotherapy (> 40 Gy) with significant areas of anticipated overlap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Koyfman, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (SBRT)
Started | 3
Completed | 2
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 84 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Head and Neck SBRT
Description: Maximum tolerated dose of SBRT in this patient population determined by the dose escalation design with doses '40Gy' and '45Gy all in 5 fractions'.
Time Frame: 3 months
Population: Patients who received treatment. MTD was not able to be determined because only three patients enrolled and no DLTs were observed. A recommended MTD could only be made if enough patients had accrued to assess toxicities in the different dosage levels.
Groups:
- Treatment (SBRT): Patients undergo Stereotactic Body Radiation Therapy in 5 fractions at least 40 hours apart over 10-18 days.
  Three dose levels: 40Gy and 45Gy all in 5 fractions. Each initial dose level will have 6 patients allocated to them. All patients are assessed at their 3 month post SBRT visit for Dose-Limiting Toxicities (DLTs). If ≤1 patient experiences a DLT, patients will be enrolled at the next dose level. If ≥3 patients experience a DLT, further accrual will be permanently halted and the study stopped. If 2 patients experience a DLT, then an additional 6 patients will be enrolled at the same dose level. In this setting, if ≤ 3/12 patients have a DLT, patients will be enrolled at the next dose level. If ≥ 4/12 patients have a DLT, further accrual will be permanently halted and the study stopped and 35 Gy will not be recommended as safe.
  The dosing strategy for the 2nd (45Gy) cohort will be identical to the first.
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 0

2. Primary Outcome: Incidence of Dose Limiting Toxicities (DLTs)
Description: Number of patients with dose limiting toxicity events graded according to CTCAE Version 4.0
Time Frame: 3 months from start of treatment
Population: Participants who enrolled in study and were treated.
Measure: Number; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimates will be used to plot overall survival - the number of patients alive at 12 months followup
Time Frame: Up to 12 months
Population: Patients who went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Local Progression Free Survival
Description: Kaplan-Meier estimates will be used to plot local progression free survival.
Time Frame: Up to 12 months
Population: No patients were alive at 12 months, so no analysis was done.
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Measured According to Standard Response Evaluation Criteria in Solid Tumors
Description: Trend tests will be used to investigate the relationship between SBRT dose and response.
Time Frame: Up to 12 months
Population: There was insufficient patient accrual to perform additional statistical analysis.
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of SBRT Related Morbidity
Description: Number of patients who experiences SBRT-related morbidity according to NCI CTCAE v 4.0
Time Frame: Up to 12 months
Population: Patients who were eligible for evaluation for SBRT-related morbidity incidence
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 1
Participants | 1

7. Secondary Outcome: Quality of Life Assessed by Functional Assessment of Cancer Therapy-Head and Neck Questionnaire
Description: Repeated analysis of variance measures will be used to analyze the quality of life data.
Time Frame: Up to 12 months
Population: No patient was able to complete 3 month follow up to provide this QOL information
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment to end of study (over a period of approximately 6 months).
Groups:
- Treatment (SBRT): Patients undergo Stereotactic Body Radiation Therapy in 5 fractions at least 40 hours apart over 10-18 days.
  Stereotactic Body Radiation Therapy: Undergo SBRT
  Positron Emission Tomography: Undergo PET/CT
  Computed Tomography: Undergo PET/CT
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Treatment (SBRT)
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SBRT) (N=3)
pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to slow accrual the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT02388932/Prot_SAP_000.pdf